CLINICAL TRIAL: NCT04759859
Title: Relationship Between Neuropsychological Functioning and Cerebral Perfusion in Patients Undergoing Carotid Endarterectomy
Brief Title: Neuropsychological Functioning and Cerebral Perfusion Post Carotid Endarterectomy
Status: Withdrawn | Type: Observational
Why Stopped: logistical issues with coordinating the clinical and testing areas
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Ali AbuRahma, Professor of Surgery, CAMC Health System
Other Study IDs: 1997246
Record Dates: First submitted 2013-11-27; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2014-01

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid Endarterectomy; Neurocognitive Functioning; Cerebral Perfusion
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Carotid Endarterectomy (CEA): 70 participants undergoing CEA
- Other Peripheral Vascular Surgery: 30 participants undergoing other peripheral vascular surgical procedures

SUMMARY:
The study aims to investigate the relationship between neuropsychological functioning and brain perfusion in patients undergoing carotid endarterectomy and control patients undergoing other peripheral vascular procedures.

DETAILED DESCRIPTION:
Carotid endarterectomy (CEA) is a vascular surgical procedure that is aimed at reducing accumulated cholesterol and fats in carotid arteries. While some research indicates that CEA is associated with improvements in neuropsychological functioning, other studies have identified deficits in neuropsychological functioning following CEA. The factors associated with these different outcomes are unclear. Identification of the factors that mediate post-CEA neuropsychological functioning outcomes may allow for the development of interventions that would improve such outcomes. Recent research has identified a relationship between post-CEA neuropsychological deficits, and cerebral blood flow in certain areas of the brain, with some indication that brain cell loss following CEA may be a key factor. The proposed study will explore changes in cerebral blood flow through the use of diffusion-weighted magnetic resonance images (DW-MRI) to investigate the relationship between neuropsychological functioning and brain perfusion in 70 CEA patients and to compare neuropsychological functioning of the CEA patients to a control group of 30 patients undergoing other peripheral vascular surgical procedures. Patients' neuropsychological functioning will be assessed pre, post and six months after the CEA or peripheral vascular surgery. Additionally DW-MRI will be assessed pre and post surgery for the patients undergoing CEA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective carotid endarterectomy or other peripheral vascular surgical procedures.
* Ages 40-90

Exclusion Criteria:

1. History of Substance Use:

   History of cocaine use within the past 12 months. Tetrahydrocannabinol use within the past 12 months.
2. Conditions that affect brain MRI/contraindications for MRI:

   Diagnosis of HIV. History of any traumatic brain injury. History or current diagnosis with any form of brain tumor. Current normal pressure hydrocephalus. Patients with any implanted metallic medical device, or non-removable metallic material in their body
3. Conditions that affect neuropsychological assessment:

   Diagnosis with Attention Deficit/Hyperactivity Disorder. Current major depressive episode. Current manic episode. Current psychotic episode. Diagnosis with any developmental disorder. Diagnosis with any form of dementia (MMSE<24). A score higher than 3 on the Modified Rankin Scale indicating a major stroke.
4. General Contraindications:

Diagnosis with or history of any medical condition that, based on reasonable clinical judgment, would clinically contraindicate the patient undergoing any of the study procedures.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients undergoing elective carotid endarterectomy and 30 patients undergoing other peripheral vascular surgical procedures
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-01-22 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
A battery of eight neuropsychological tests | 7 days before surgery, 1-7 days after surgery and 6 months after surgery

SECONDARY OUTCOMES:
Diffusion Weighted Magnetic Resonance Imaging | 7 days before surgery, 1-7 days after surgery

OTHER OUTCOMES:
Short Form-36 | 7 days before surgery, 1-7 days after surgery and 6 months follow-up
Beck Depression Inventory II | 7 days before surgery, 1-7 days after surgery and 6 months after surgery
State-Trait Anxiety Inventory | 7 days before surgery, 1-7 days after surgery and 6 months after surgery
An 11-point Numeric Pain Intensity Scale | 7 days before surgery, 1-7 days after surgery and 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ali AbuRahma, MD, Principal Investigator — Charleston Area Medical Center Vascular Center of Excellence
Locations (1):
- Charleston Area Medical Center Vascular Center of Excellence, Charleston, West Virginia, United States